CLINICAL TRIAL: NCT02473965
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of lGIV-C as a Corticosteroid Sparing Agent in Corticosteroid Dependent Patients With Generalized Myasthenia Gravis
Brief Title: Efficacy and Safety of IGIV-C in Corticosteroid Dependent Patients With Generalized Myasthenia Gravis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GTI1306
Record Dates: First submitted 2015-06-14; First posted 2015-06-17 (Estimated); Results first posted 2020-02-26 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- IGIV-C (Experimental): An IGIV-C loading dose of 2 g/kg and maintenance dose of 1 g/kg will be administered in CS dependent subjects with MG.
  Interventions: Drug: IGIV-C
- Placebo (Placebo Comparator): 0.9% sodium chloride injection, USP or equivalent
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IGIV-C — Run-Phase: 1 loading dose of 2 g/kg IGIV-C and 2 maintenance doses of 1 g/kg IGIV-C
  Corticosteroid Tapering/IGIV-C Maintenance Phase: 1 g/kg IGIV-C every 3 weeks for up to 36 weeks
  Arms: IGIV-C
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of Immune Globulin (Human), 10% Caprylate/Chromatography Purified (IGIV-C) as a corticosteroid (CS)-sparing agent in subjects with CS-dependent Myasthenia Gravis (MG).

DETAILED DESCRIPTION:
This study consists of 2 phases: IGIV-C Run-in Phase and Corticosteroid Tapering/IGIV-C Maintenance Phase.

In the Run-in Phase, subjects will receive a total of 3 doses of IGIV-C (1 loading dose of 2 g/kg and 2 maintenance doses of 1 g/kg) while maintaining a stable dose of corticosteroids.

In the CS Tapering/IGIV-C Maintenance Phase, subjects will continue 1 g/kg IGIV-C and begin a prescribed CS tapering regimen where the CS dose is decreased every 3 weeks.

Approximately 60 subjects are planned to be enrolled in the study across multiple centers in North America and Europe. The total duration of study participation for each subject is up to 45 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Anti-acetylcholine receptor antibody positive
* Confirmed diagnosis of generalized MG historically meeting the clinical criteria for diagnosis of MG defined by the Myasthenia Gravis Foundation of America (MGFA) classification of Class II, III, IV, or V historically
* At Screening, subjects may have symptoms controlled by CS or were MGFA Class II-IVa inclusive (Class IVb and Class V excluded). Subjects who only have a history of ocular MG may not enroll.
* On systemic CS for a minimum period of at least 3 months and on a stable CS dose of >=15 mg/day and <=60 mg/day (prednisone equivalent) for the month prior to Screening.
* Had a tapering CS dose that the study investigator considered to be appropriate.
* At least 1 previous completed attempt to taper CS in order to minimize CS dose (lowest feasible dose based on observed MG signs and symptoms)

Exclusion Criteria:

* Any dose change in concomitant immunosuppressant therapy, other than CS, in the prior 6 months
* Any change in CS dose or acetylcholinesterase inhibitor (e.g., pyridostigmine) dose in the 1 month prior to Screening
* A 3-point change in Quantitative Myasthenia Gravis score, increased or decreased, between the Screening/Week -3 (Visit 0) and Baseline (Week 0 [Visit 1])
* Any episode of myasthenic crisis (MC) in the 1 month prior to Screening, or (at any time in the past) MC or hospitalization for MG exacerbation associated with a previous CS taper attempt
* Evidence of malignancy within the past 5 years (non-melanoma skin cancer, carcinoma in situ of cervix is allowed) or thymoma potentially requiring surgical intervention during the course of the trial (intent to perform thymectomy)
* Thymectomy within the preceding 6 months prior to Screening
* Rituximab, belimumab, eculizumab or any monoclonal antibody used for immunomodulation within the past 12 months prior to Screening
* Have received immune globulin treatment given by IV, subcutaneous, or intramuscular route within the last 3 months prior to Screening
* Received plasma exchange performed within the last 3 months prior to Screening
* History of anaphylactic reactions or severe reactions to any blood-derived product
* History of recent (within the last year) myocardial infarction or stroke
* Uncontrolled congestive heart failure; embolism; or historically documented (within the last year) electrocardiogram changes indicative of myocardial ischemia or atrial fibrillation
* Current known hyperviscosity or hypercoagulable state
* Currently receiving anti-coagulation therapy. Oral anti-platelet agents are allowed (e.g., aspirin, clopidogrel, ticlopidine)
* Females of child-bearing potential who are pregnant, have a positive serum pregnancy test, breastfeeding, or are unwilling to practice a highly effective method of contraception throughout the study.
* Renal impairment
* Aspartate aminotransferase or alanine aminotransferase levels exceeding more than 2.5 times the upper limit of normal for the expected normal range for the testing laboratory.
* Hemoglobin (Hb) levels <9 g/dL

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-06; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (39):
- United States (14):
  - University of California-Irvine, Orange, California
  - Yale University School of Medicine, Department of Neurology, New Haven, Connecticut
  - University of Florida at Shands Jacksonville, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - Georgia Regents University, Augusta, Georgia
  - Indiana University, Indianapolis, Indiana
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Columbia University Medical Center, New York, New York
  - Ohio State University Wexner Medical Center, Neurology Department, Columbus, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Houston Methodist Neurological Institute, Houston, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Washington Medical Center, Seattle, Washington
- UZ Leuven, Leuven, Belgium
- Canada (2):
  - London Health Sciences Centre- University Hospital, London, Ontario
  - University Health Network (UHN) - Toronto General Hospital, Toronto, Ontario
- Czechia (3):
  - Fakultni nemocnice Brno, Dept of Neurologicka klinika, Brno
  - Fakultni nemocnice Ostrava, Ostrava - Poruba
  - Vseobecna fakultni nemocnice v Praze, Dept of Neurologicka klinika, Prague
- East Tallinn Central Hospital, Tallinn, Estonia
- France (2):
  - CHU Strasbourg - Nouvel Hôpital Civil, Clinique Neurologique, Strasbourg, Bas Rhin
  - CHU de Toulouse - Hôpital Purpan, Service de Neurologie Générale, Toulouse, Haute Garonne
- Germany (8):
  - Universitaetsklinikum Regensburg, Parent, Regensburg, Bavaria
  - Universitaetsklinikum Giessen und Marburg GmbH Standort Marburg, Marburg, Hesse
  - Universitaetsmedizin Goettingen, Parent, Göttingen, Lower Saxony
  - Fachkrankenhaus Hubertusburg gGmbH, Klinik f. Neurologie, Wermsdorf, Saxony
  - Krankenhaus Martha-Maria Halle-Doelau, Klinik fuer Neurologie, Halle, Saxony-Anhalt
  - Universitaetsklinikum Jena, Klinik fuer Neurologie, Jena, Thuringia
  - Charité Universitaetsmedizin Berlin, Klinik für Neurologie, Berlin
  - Universitaetsklinikum Hamburg-Eppendorf, Klinik und Poliklinik, Hamburg
- Hungary (3):
  - Jahn Ferenc Del-pesti Korhaz es Rendelointezet, Neurologiai Osztaly, Budapest
  - Pest Megyei Flor Ferenc Korhaz, Neurologia es Stroke Osztaly, Kistarcsa
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged
- Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas, Lithuania
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Dept of Neurology, Gdansk
  - Krakowska Akademia Neurologii Sp z o.o. Centrum Neurologii Klinicznej, Krakow
  - III Szpital Miejski w Lodzi im. Dr K. Jonschera, Lodz
  - Samodzielny Publiczny Centralny Szpital Kliniczny, Warsaw

REFERENCES:
- [Derived] Bril V, Szczudlik A, Vaitkus A, Rozsa C, Kostera-Pruszczyk A, Hon P, Bednarik J, Tyblova M, Kohler W, Toomsoo T, Nowak RJ, Mozaffar T, Freimer ML, Nicolle MW, Magnus T, Pulley MT, Rivner M, Dimachkie MM, Distad BJ, Pascuzzi RM, Babiar D, Lin J, Querolt Coll M, Griffin R, Mondou E. Randomized Double-Blind Placebo-Controlled Trial of the Corticosteroid-Sparing Effects of Immunoglobulin in Myasthenia Gravis. Neurology. 2023 Feb 14;100(7):e671-e682. doi: 10.1212/WNL.0000000000201501. Epub 2022 Oct 21. PMID 36270895
- [Derived] Dalakas MC, Meisel A. Immunomodulatory effects and clinical benefits of intravenous immunoglobulin in myasthenia gravis. Expert Rev Neurother. 2022 Apr;22(4):313-318. doi: 10.1080/14737175.2022.2057223. Epub 2022 Apr 5. PMID 35350948

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty subjects with a confirmed diagnosis of generalized myasthenia gravis (MG) historically meeting the clinical criteria for MG diagnosis Class II, III, IV or V of the Myasthenia Gravis Foundation of America were randomized. The study was conducted in 8 countries from November 2015 to February 2019.
Pre-assignment Details: Subjects had symptoms at screening controlled by corticosteroids (CS), had been dependent on systemic CS for at least the preceding 3 months and had received a stable dose of CS for at least 1 month immediately prior to the screening visit.
Groups:
- IGIV-C: Investigational Product (IP) Run-in Maintenance Phase (Weeks 0-9): Subjects randomized to receive Immune Globulin (Human), 10% Caprylate/Chromatography Purified (IGIV-C) were given a loading dose of 2 grams per kilogram (g/kg) by intravenous (IV) infusion at Baseline/Week 0 (Visit 1) and 2 maintenance doses of 1 g/kg at Weeks 3 and 6 (Visits 2 and 3). The CS dose remained stable in this phase.
  CS Tapering/IP Maintenance Phase (Weeks 9-36): Subjects continued to receive maintenance doses (1 g/kg) every third week from Week 9 (Visit 4) up to Week 36 (Visit 13). Prescribed CS tapering began at Week 9 (Visit 4) after the third maintenance dose of IGIV-C was given. The last CS dose reduction was at Week 36 (Visit 13).
  Safety/Follow-up Phase: Follow-up visits were at Weeks 39, 42 and 45 (Visits 14, 15 and 16). If considered medically indicated, the investigator could increase the CS dose after the Week 39 (Visit 14) assessments.
- Placebo: IP Run-in Maintenance Phase (Weeks 0-9): Subjects randomized to receive placebo were given 3 doses of placebo matching IGIV-C by IV infusion at Baseline/Week 0 (Visit 1) and at Weeks 3 and 6 (Visits 2 and 3). The CS dose remained stable in this phase.
  CS Tapering/IP Maintenance Phase (Weeks 9-36): Subjects continued to receive maintenance doses of placebo matching IGIV-C every third week from Week 9 (Visit 4) up to Week 36 (Visit 13). Prescribed CS tapering began at Week 9 (Visit 4) after the third maintenance dose of placebo was given. The last CS dose reduction was at Week 36 (Visit 13).
  Safety/Follow-up Phase: Follow-up visits were at Weeks 39, 42 and 45 (Visits 14, 15 and 16). If considered medically indicated, the investigator could increase the CS dose after the Week 39 (Visit 14) assessments.
Period: Overall Study
Arm/Group | IGIV-C | Placebo
Started | 30 | 30
Completed (Completed up to Week 45) | 18 | 20
Not Completed | 12 | 10
Not completed — Adverse Event | 6 | 4
Not completed — MG worsening | 4 | 1
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Population: The modified intent-to-treat (mITT) population included all randomized subjects who received at least 1 dose of study medication. Subjects were classified according to randomized treatment.
Groups:
- IGIV-C: IP Run-in Maintenance Phase (Weeks 0-9): Subjects randomized to receive IGIV-C were given a loading dose of 2 g/kg by IV infusion at Baseline/Week 0 (Visit 1) and 2 maintenance doses of 1 g/kg at Weeks 3 and 6 (Visits 2 and 3). The CS dose remained stable in this phase.
  CS Tapering/IP Maintenance Phase (Weeks 9-36): Subjects continued to receive maintenance doses (1 g/kg) every third week from Week 9 (Visit 4) up to Week 36 (Visit 13). Prescribed CS tapering began at Week 9 (Visit 4) after the third maintenance dose of IGIV-C was given. The last CS dose reduction was at Week 36 (Visit 13).
  Safety/Follow-up Phase: Follow-up visits were at Weeks 39, 42 and 45 (Visits 14, 15 and 16). If considered medically indicated, the investigator could increase the CS dose after the Week 39 (Visit 14) assessments.
Arm/Group | IGIV-C | Placebo | Total Title
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (16.99) | 48.5 (14.51) | 48.1 (15.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 34
  Male | 14 | 12 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 30 | 28 | 58
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 27 | 27 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Baseline Daily Prednisone Equivalent Dose Level Stratification Categories [Count of Participants; unit: Participants]
  15 mg to 40 mg/day | 29 | 28 | 57
  41 to 60 mg/day | 1 | 2 | 3
Baseline QMG Total Score [Mean (Standard Deviation); unit: units on a scale] — The Quantitative Myasthenia Gravis (QMG) total score was the sum of the 13 items used to measure spirometry and muscle strength and ranges from 0 to 39 (higher values indicate greater severity of illness). The QMG total scores were used to assess MG worsening.
  units on a scale | 12.1 (6.98) | 11.2 (6.48) | 11.6 (6.69)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects Achieving a 50% or Greater Reduction in CS Dose (Prednisone or Equivalent) From Baseline to Week 39
Description: The average daily CS dose was derived for each subject at each scheduled visit based on the prescribed dose and the time interval taking into account any prescribed dose changes between routinely scheduled visits. Subjects who discontinued the study early with adverse outcomes related to MG were considered as not achieving a 50% or greater reduction. The missing dose reduction at Week 39 was imputed using the worst observation carried forward (WOCF) method. For subjects who did not have CS dose prescribed at Week 39 due to other reasons, the last observation carried forward (LOCF) method was used to impute the prescribed CS dose at Week 39. Baseline was defined as the last non-missing measurement taken prior to first dose of study medication. The percent of subjects achieving ≥50% reduction in CS dose from baseline to Week 39 is presented for each treatment group overall and for the baseline daily prednisone equivalent dose level stratification categories.
Time Frame: Baseline/Week 0 (Visit 1) and Week 39 (Visit 14).
Population: The mITT population included all randomized subjects who received at least 1 dose of study medication. Subjects were classified according to randomized treatment.
Measure: Number; unit: percentage of subjects
Arm/Group | IGIV-C | Placebo
Number analyzed (Participants) | 30 | 30
percentage of subjects
  All subjects | 60.0 | 63.3
  15 mg to 40 mg/day: number analyzed (Participants) | 29 | 28
  15 mg to 40 mg/day | 58.6 | 60.7
  41 mg to 60 mg/day: number analyzed (Participants) | 1 | 2
  41 mg to 60 mg/day | 100.0 | 100.0
Statistical Analysis 1: Comparison: IGIV-C vs Placebo; An unstratified analysis using Fisher's exact test was used for treatment comparison without adjustment for stratified baseline prednisone equivalent dose level due to the small cell size. The odds ratio and confidence intervals are calculated overall (i.e. all mITT subjects); Test type: Superiority; p = 1.00, Fisher Exact — The statistical inference was tested as 2-sided with alpha=0.05; Odds Ratio (OR) = 0.868, 95% CI 2-sided [0.270 to 2.787]

2. Secondary Outcome: Mean Percent Change in Daily CS Dose (Prednisone or Equivalent) From Baseline to Week 39
Description: The average daily CS dose was derived for each subject at each scheduled visit based on the prescribed dose and the time interval taking into account any prescribed dose changes between routinely scheduled visits. For subjects who discontinued the study early with adverse outcomes related to MG, the missing dose reduction at Week 39 was imputed using the WOCF method. For subjects who had missing CS dose reduction at Week 39 due to other reasons, the missing CS dose was imputed using the LOCF method. Baseline was defined as the last non-missing measurement taken prior to first dose of study medication. The least squares (LS) mean percent change from baseline in daily CS dose to Week 39 is presented for each treatment group.
Time Frame: Baseline/Week 0 (Visit 1) and Week 39 (Visit 14).
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | IGIV-C | Placebo
Number analyzed (Participants) | 30 | 30
percent change | -52.57 (8.835) | -54.15 (8.835)
Statistical Analysis 1: Comparison: IGIV-C vs Placebo; Treatment comparison of percent change in daily CS dose from baseline to Week 39. The Analysis of Covariance model included the percent change from baseline in daily CS dose as the dependent variable, treatment as a fixed effect and baseline daily CS dose as covariate; Test type: Superiority; p = 0.900, ANCOVA; LS mean difference = 1.58, 95% CI 2-sided [-23.52 to 26.68], Standard Error of Mean 12.536

3. Secondary Outcome: Median Time to First Episode of MG Worsening
Description: The time to the first episode of MG worsening was defined as the time between baseline and the first instance of QMG total score increase by ≥4 points relative to Baseline/Week 0. The QMG total score is the sum of all 13 items and ranges from 0 to 39. Higher values represent greater severity of illness. If one or more items were missing at a given assessment, the total score was set to missing. The median time to MG worsening was calculated based on Kaplan-Meier methodology. Baseline was defined as the last non-missing measurement taken prior to the first dose of study medication.
Time Frame: From Baseline/Week 0 (Visit 1) to Week 39 (Visit 14).
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | IGIV-C | Placebo
Number analyzed (Participants) | 30 | 30
weeks | NA [33.10 to NA] — The median and 75th percentile were non-estimable as >50% of subjects did not have an episode of MG worsening. | NA [30.10 to NA] — The median and 75th percentile were non-estimable as >50% of subjects did not have an episode of MG worsening.

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAEs) were collected from Baseline/Week 0 to Week 39 (approximately 9 months).
Description: TEAEs are presented for the Safety population which consisted of all randomized subjects who received any amount of study medication. Subjects were classified according to the treatment received.
Arm/Group | IGIV-C | Placebo
All-Cause Mortality (participants affected / at risk) | 1/30 | 2/30
Serious Adverse Events (participants affected / at risk) | 4/30 | 6/30
Other Adverse Events (participants affected / at risk) | 21/30 | 24/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IGIV-C (N=30) | Placebo (N=30)
Myasthenia gravis (Nervous system disorders) | 4 (4) | 1 (1)
Myasthenia gravis crisis (Nervous system disorders) | 1 (1) | 2 (2)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IGIV-C (N=30) | Placebo (N=30)
Headache (Nervous system disorders) | 10 (15) | 3 (3)
Myasthenia gravis (Nervous system disorders) | 7 (7) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 6 (7) | 3 (3)
Nausea (Gastrointestinal disorders) | 5 (6) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 2 (2) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Blood pressure increased (Investigations) | 2 (5) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (3)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2) | 5 (6)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 3 (4)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Red blood cell count decreased (Investigations) | 2 (3) | 0 (0)
Viral infection (Infections and infestations) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3) | 0 (0)
White blood cell count decreased (Investigations) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (6)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/65/NCT02473965/SAP_000.pdf
  • Study Protocol (2016-12-23): https://cdn.clinicaltrials.gov/large-docs/65/NCT02473965/Prot_001.pdf